CLINICAL TRIAL: NCT05768009
Title: Respiratory and Analgesic Effects of Interscalene Block Versus Pericapsular Nerve Block and Superficial Cervical Plexus Block for Arthroscopic Shoulder Surgery
Brief Title: Interscalene Block Versus Pericapsular Nerve Block and Superficial Cervical Plexus Block for Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principle Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Interscalene block
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Interscalene Block; Superficial Cervical Block
Keywords: Interscalene , Pericapsular Nerve Block , Superficial Cervical Plexus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene brachial plexus block (ISB) (Experimental): • Group A will include 21 patients who will undergo the procedure under general anesthesia and ultrasound guided Interscalene brachial plexus block using 10 ml bupivacaine 0.25%.the interscalene block will be performed when the patient is in a supine position, with his/her head slightly elevated and turned away from the side to be blocked. The linear ultrasound probe (frequency 10-15 MHz) will be used with the depth setting of 2-4 cm. The probe will be initially placed near the midline of clavicle at the level of cricoid cartilage and scanned laterally to identify the carotid artery and internal jugular vein underneath the sternocleidomastoid muscle. By moving the probe laterally, the anterior scalene muscle will be identified below the lateral edge of the sternocleidomastoid. A groove containing the hypoechoic nerve structures will usually be identified. 10 mL of 0.25 bupivacaine will be injected into scalene groove around the nerve roots.
  Interventions: Procedure: Interscalene brachial plexus block (ISB)
- pericapsular nerve block and superficial cervical plexus blocks (Experimental): • Group B will include 21 patients who will undergo the procedure under general anesthesia and combined pericapsular nerve block and superficial cervical plexus blocks (using 10 and 5 ml bupivacaine 0.25% respectively).
  the patient's arm will be placed in external rotation and abducted at 45 degrees. The linear ultrasound probe will be placed longitudinally between the coracoid process and the humeral head. After identification of the humeral head, the subscapularis tendon and the deltoid muscle over it, a 50-mm sonovisible needle will be inserted using the "in plane" technique. The needle tip will be placed between the deltoid muscle and subscapularis tendon, and 10 ml of 0.25% bupivacaine will be injected.
  Interventions: Procedure: Interscalene brachial plexus block (ISB)

INTERVENTIONS:
Procedure: Interscalene brachial plexus block (ISB) — • Group A will include 21 patients who will undergo the procedure under general anesthesia and ultrasound guided ISB using 10 ml bupivacaine 0.25%.

SUMMARY:
Interscalene brachial plexus block (ISB) is considered the standard nerve block for shoulder surgery . It provides superior analgesia and reduced opioid-related adverse effects . However, it is challenging to perform and may be associated with a high incidence of ipsilateral hemidiaphragmatic paresis, resulting from a phrenic nerve block . Although that complication could be decreased with modified local anesthetic dosing and ultrasound-guided needle placement , its incidence significantly impair the mechanics of breathing leading to postoperative morbidity, making that block undesirable in patients with impaired pulmonary functions .

This clinical problem has recently received considerable attention, with several calls to seek alternatives to interscalene block in shoulder arthroscopy [18]. So, the need for a safer ISB alternative has prompted researchers to examine several options, including but not limited to the suprascapular [19] and pericapsular nerve blocks .

Pericapsular nerve block has been studied extensively in hip surgeries , and some physicians suggested that it can be safely applied for analgesia and can be part of surgical anesthesia in shoulder arthroscopic surgery. It induces blockade of the articular branches that innervate the glenohumeral joint . The block of this area does not cause motor block or pulmonary complications, nor result in muscle laxity, blocking only the shoulder and the upper third of the humerus .

The cervical plexus is formed by the ventral rami of C1-C4 cervical roots. It can be blocked at the superficial, intermediate and at the deep level [24]. The superficial cervical plexus block results in anesthesia of skin over the anterolateral neck, skin overlying the clavicle and the sternoclavicular joint, anterior and retroauricular areas . Although that block is effective in pain management after surgeries involving the distal clavicle, it has been poorly described in shoulder arthroscopy.

DETAILED DESCRIPTION:
Study design

* This is a prospective randomized trial. Setting
* Anesthesiology and Pain Management Department, Tanta University Hospitals, Orthopedic Department, Tanta, Egypt.

Study duration

• The study will be conducted over a six-month duration, starting from April 2023 till the end of October 2023.

Study participants

* A total of 42 patients will be included in our study. Method of randomization
* Randomization will be performed via the "sealed envelope" method. Patient consent
* All patients will sign an informed written consent after explaining the benefits and possible complications of each regional block approach.

Study groups The included patients will be randomly assigned into two equal groups;

* Group A will include 21 patients who will undergo the procedure under general anesthesia and ultrasound guided ISB using 10 ml bupivacaine 0.25%.
* Group B will include 21 patients who will undergo the procedure under general anesthesia and combined pericapsular nerve block and superficial cervical plexus blocks (using 10 and 5 ml bupivacaine 0.25% respectively).

Inclusion criteria

* Adult patients aged between 18 and 65 years.
* Classification as class I or II according to the American Society of Anesthesiologists (ASA).
* Patients scheduled for elective arthroscopic shoulder procedures. Patient evaluation
* All patients will be subjected to detailed history taking, clinical examination, radiological shoulder assessment, in addition to routine preoperative laboratory investigations.
* All patients will be also assessed by the anesthetist prior to admission and classified according to the ASA classification.
* Patients will be also taught how to express their pain via an eleven-point scale (numerical rating scale or NRS), ranging from 0 to 10, with 0 for no pain at all, and 10 for the worst pain ever.

Breathing Assessments After consent and randomization, and before block performance, all patients will have baseline diaphragmatic excursion and pulmonary function testing. Diaphragmatic excursion with shallow (sniff) and deep (sigh) breathing will be evaluated using a low-frequency ultrasound transducer (Mindray machine, China) in M-mode with patients in the sitting position, as previously described by Cuvillon . Patients will be scanned using a low intercostal or subcostal view using the liver or spleen as an acoustic window. Patients will be informed to inhale deeply and exhale completely (sigh breath), and an image will be taken. M-mode was used to evaluate the excursion distance. These measurements will be then used to determine level of diaphragmatic paralysis as defined by Renes , with no paralysis 0 to 25% (percent change from baseline), partial paralysis 25 to 75%, and complete paralysis 75% or greater. This will be repeated with the patient taking a sniff breath, a quick short inhalation through the nose with a closed mouth. Each measurement will be performed twice, and the values will be averaged. Diaphragm movement will be measured in centimetres Assessment of pulmonary function tests will be done when the patient is in the sitting position using a hand-held spirometer. It will be used to measure forced vital capacity, FEV1, FEV1/forced vital capacity ratio, and flow rate in liters per second. Three separate measurements will be taken and averaged for each patient. Identical breathing assessments will be repeated postoperatively at two time points:30 min after emergence from anesthesia in the postanesthesia care unit (PACU), and 24 h after block placement with the patient on the surgical ward. pulmonary function test and diaphragmatic excursion will be evaluated by another anesthesiologist who is blinded for the groups.

Preoperative care

* A peripheral IV line will be secured into a suitable forearm vein (on the upper limb contralateral to the surgery side). Basic hemodynamic monitoring including pulse oximetry, noninvasive blood pressure, heart rate and electrocardiogram will be connected to all patients.
* All patients will receive 2 mg midazolam and 50 mcg fentanyl on arrival to the operating room.

The block procedure All blocks will be performed by Ultrasound machine (Phillips®, Cx-50, Amsterdam, Netherlands) with a Superficial probe 5-12 MHz will be used in the two groups under complete aseptic condition after proper skin draping. Anesthesiologist who will make the ultrasound nerve blocks has no any other role in the study .

criteria are fulfilled. Postoperative assessment

* After the end of the arthroscopic intervention, all patients will be transferred to the PACU then to the internal ward, where close monitoring will be done. Hemodynamic Parameters: (MAP & HR) will be recorded before block performance, intraoperatively at 15 & 30 minutes after block and, then every 30 min till the end of surgery, and before discharge from PACU, then at 2,4,6,12,18,24 hours postoperative.
* The same diaphragmatic ultrasound measurements and spirometry will be performed at PACU 30 min postoperative then 24 hours after the operation.
* Postoperative pain will be assessed via the NRS, and its values will be recorded at PACU and then at, 2, 4, 6, 12, 18, 24 h after arthroscopy.
* Analgesia will be achieved by IV acetaminophen (1 gm/8 hours) in addition to IV ketorolac (30 mg/12 hours. If the patient reports a breakthrough pain (NRS > 4), the patient will be given intravenous morphine (Sunny pharmaceutical, Egypt) as rescue analgesia in a dose 0.05mg/kg.
* The duration till the first breakthrough pain and the total morphine consumption will be recorded.
* Patient satisfaction with the pain management intervention will be graded as 4 point Likert scale, from 0 to 4, as follows; weak, medium, good, very good and excellent, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 65 years, Classification as class I or II according to the American Society of Anesthesiologists (ASA) , Patients scheduled for elective arthroscopic shoulder procedures.

Exclusion Criteria:

* • Age beyond the previous limits.

  * Refusal to participate in the study.
  * Patients with peripheral neuropathy.
  * Patients with chronic chest diseases affecting their pulmonary function results.
  * ASA class > II.
  * Bleeding diathesis.
  * Pregnancy.
  * Recent history of anticoagulant or antiplatelet drug intake.
  * Cutaneous infection at the injection site.
  * Patients with pacemakers.
  * Patients with AV block.
  * Known allergy to local anesthetics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-25 (Estimated); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
• The incidence of postoperative diaphragmatic paralysis | 24 hour
  The same diaphragmatic ultrasound measurements will be performed at PACU 30 minutes postoperative then 24 hours after the operation

SECONDARY OUTCOMES:
• Postoperative pain will be assessed via the NRS, and its values will be recorded at PACU and then at, 2, 4, 6, 12, 18, 24 hour after arthroscopy. | 24 hour
  • Postoperative pain will be assessed via the NRS, and its values will be recorded at PACU and then at, 2, 4, 6, 12, 18, 24 hour after arthroscopy.
The total amount of analgesia and 1st rescue analgesia | 24 hour
  • The duration till the first breakthrough pain and the total morphine consumption will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ELgharbiaa, Egypt